CLINICAL TRIAL: NCT02647944
Title: Pilot Study of the Effect of Liraglutide on Weight Loss and Gastric Functions in Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Michael Camilleri, Principle Investigator, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 15-001783; R56DK067071 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2015-12-31; First posted 2016-01-06 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liraglutide (Active Comparator): Saxenda initiated at 0.6mg S.C. daily for 1 week; subjects will return to the Clinical Research Unit (CRU) each week until an increase by 0.6 mg/day in weekly intervals to a dose of 3.0 mg/day is achieved. Once maintenance dose of 3.0 mg is achieved, subjects will return approximately every 4 weeks to obtain new supply of study medication.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo initiated at 0.6mg S.C. daily for 1 week; subjects will return to the Clinical Research Unit (CRU) each week until an increase by 0.6 mg/day in weekly intervals to a dose of 3.0 mg/day is achieved. Once maintenance dose of 3.0 mg is achieved, subjects will return approximately every 4 weeks to obtain new supply of study medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Initiate at 0.6mg S.C. daily for 1 week; subjects will return to the Clinical Research Unit (CRU) each week until an increase by 0.6mg/day in weekly intervals to a dose of 3.0 mg/day is achieved (~4 weeks). Once maintenance dose of 3.0 mg is achieved, subjects will return approximately every 4 weeks to obtain new supply of study medication.
  Other Names: Saxenda
  Arms: Liraglutide
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study was being done to assess the stomach emptying effect of a maximum dose of 3 mg Liraglutide compared to placebo in subjects who are overweight or obese. Liraglutide is a medication approved by the Food and Drug Administration (FDA) for routine clinical use.

DETAILED DESCRIPTION:
The objective of this study was to compare effects of liraglutide and placebo over 16 weeks on gastric motor functions, satiation, satiety and weight in obese patients. Subjects were randomized to liraglutide or placebo. Liraglutide or placebo was escalated by 0.6mg/day each week for 5 weeks and continued until week 16. At baseline and after 16 weeks' treatment, the investigators measured weight, gastric emptying of solids (GES), gastric volumes, satiation (maximum tolerated volume of liquid nutrient drink), and satiety. GES was also measured at 5 weeks.

During the study, the subjects received standardized dietetic and behavioral advice for weight reduction therapy. All subjects were given a standard text for information and met with a behavioral psychologist who has expertise in obesity treatment at the baseline visit and at visits at weeks 4,8, and 12. Additionally, the subjects had brief contact with a member of the study team every 4 weeks to inquire about their adherence to study protocol, any difficulties they were experiencing, whether they were reading their text assignments, and to answer any additional questions.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese adults (≥30 kg/m^2 or ≥27 kg/m^2 with an obesity-related co-morbidity).
* Subjects residing within 125 miles of Mayo Clinic in Rochester, Minnesota.
* Healthy individuals with no unstable psychiatric disease and not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, or endocrine (other than hyperglycemia type 2 diabetes mellitus on metformin) disorders.
* Women of childbearing potential will be using an effective form of contraception, and have negative pregnancy tests within 48 hours of enrolment and before each radiation exposure.
* Subjects must have the ability to provide informed consent before any trial-related activities.

Exclusion criteria:

* Weight exceeding 137 kilograms (safety limit of camera for measuring gastric volumes).
* Abdominal surgery other than appendectomy, Caesarian section or tubal ligation.
* Positive history of chronic gastrointestinal diseases, systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., orlistat.
* Patients with a personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia-type 2.
* Patients with a personal history of pancreatitis (acute or chronic)
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory, a self-administered alcoholism screening test (AUDIT-C), and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a Hospital Anxiety Depression (HAD) score >8 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Intake of medication, whether prescribed or over the counter (except multivitamins), within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, thyroxin replacement therapy and any medication administered for co-morbidities as long as they do not alter gastrointestinal motility including gastric emptying (GE) and gastric accommodation. For example, statins for hyperlipidemia, diuretics, β-adrenergic blockers,Angiotensin Converting Enzyme (ACE) inhibitors and angiotensin antagonists for hypertension, and metformin for type 2 diabetes mellitus or prediabetes are permissible. In contrast, resin sequestrants for hyperlipidemia [which may reduce GE and reduce appetite, α2-adrenergic agonists for hypertension, or other glucagon-like peptide-1 receptor agonists (GLP-1) receptor agonists (exenatide) or amylin analogs (pramlintide) are not permissible because they significantly affect GE and/or gastric accommodation.
* Hypersensitivity to the study medication, liraglutide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Halawi H, Khemani D, Eckert D, O'Neill J, Kadouh H, Grothe K, Clark MM, Burton DD, Vella A, Acosta A, Zinsmeister AR, Camilleri M. Effects of liraglutide on weight, satiation, and gastric functions in obesity: a randomised, placebo-controlled pilot trial. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):890-899. doi: 10.1016/S2468-1253(17)30285-6. Epub 2017 Sep 27. PMID 28958851
- [Derived] Maselli D, Atieh J, Clark MM, Eckert D, Taylor A, Carlson P, Burton DD, Busciglio I, Harmsen WS, Vella A, Acosta A, Camilleri M. Effects of liraglutide on gastrointestinal functions and weight in obesity: A randomized clinical and pharmacogenomic trial. Obesity (Silver Spring). 2022 Aug;30(8):1608-1620. doi: 10.1002/oby.23481. PMID 35894080
- [Derived] Kadouh H, Chedid V, Halawi H, Burton DD, Clark MM, Khemani D, Vella A, Acosta A, Camilleri M. GLP-1 Analog Modulates Appetite, Taste Preference, Gut Hormones, and Regional Body Fat Stores in Adults with Obesity. J Clin Endocrinol Metab. 2020 May 1;105(5):1552-63. doi: 10.1210/clinem/dgz140. PMID 31665455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between December 18, 2015 and September 1, 2016 at the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 19 | 21
Completed | 17 | 18
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.95 (11.08) | 37.81 (12.14) | 39.30 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 17 | 19 | 36
  Asian | 1 | 0 | 1
  Hispanic or Latino | 0 | 2 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40
Body Mass Index (BMI) [Mean (Inter-Quartile Range); unit: kg/m^2] | 37.2 [33.6 to 41.0] | 34.6 [33.4 to 38.9] | 36.65 [33.5 to 39.5]
Body Weight [Mean (Inter-Quartile Range); unit: kg] — Population: Body weight was not recorded at baseline for one participant in the placebo group.
  kg
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 103.7 [90.0 to 112.2] | 99.1 [90.1 to 111.2] | 103 [90.0 to 111.5]

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying of Solids Half-time (T1/2) at 5 Weeks
Description: Gastric emptying of solids was assessed by scintigraphy using a 320 Kcal 99mTc-radiolabeled egg, solid-liquid meal. Gastric Emptying Half-time was the linear interpretation of time to when 50% of radiolabeled meal emptied from the stomach.
Time Frame: 5 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
minutes | 180 [162 to 295] | 117 [96 to 137]

2. Primary Outcome: Gastric Emptying of Solids Half-time (T1/2) at 16 Weeks
Description: as for outcome 1
Time Frame: 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
minutes | 142 [120 to 177] | 113 [101 to 133]

3. Secondary Outcome: Weight Change at 5 Weeks
Description: Body weight in kg was measured at 5 weeks and compared to baseline.
Time Frame: baseline, 5 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
kg | 3.70 [2.80 to 4.80] | 0.60 [-0.30 to 1.4]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Weight Change at 16 Weeks
Description: Body weight in kg was measured at 16 weeks and compared to baseline.
Time Frame: baseline, 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
kg | 5.30 [5.20 to 6.80] | 2.5 [0.1 to 4.2]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Satiety by Buffet Meal, Total Calories Ingested at 16 Weeks
Description: Satiety (a measure of appetite) was appraised by "free feeding" buffet meal consisting of standard foods of known nutrient composition. The total amount of food consumed was analyzed by the study dietitian.
Time Frame: 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
kcal | 554.0 [406 to 687] | 680.5 [513 to 1002]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Satiation Volume to Fullness at 16 Weeks
Description: After drinking Ensure, participants recorded their sensations every 5 minutes using a numerical scale from 0 to 5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation).
Time Frame: 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
mL | 360 [360 to 600] | 600 [480 to 720]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.069, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Satiation Maximum Tolerated Volume at 16 Weeks
Description: as for outcome 6
Time Frame: 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
mL | 750 [651 to 908] | 1126 [944 to 1185]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.054, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Gastric Fasting Volume at 16 Weeks
Description: Gastric fasting volume was measured by single photon emission computed tomography (SPECT) imaging of the stomach after intravenous injection of 99mTC-pertechnetate, which is taken up by the gastric mucosa.
Time Frame: 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
mL | 231 [192 to 277] | 192 [179 to 223]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Gastric Postprandial Volume at 16 Weeks
Description: as for outcome 8
Time Frame: 16 weeks
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
mL | 705 [633 to 744] | 668 [605 to 794]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Gastric Accommodation Volume at 16 Weeks
Description: Change between postprandial and fasting whole gastric volume by 99mTc-SPECT Imaging. A noninvasive SPECT method was used to measure gastric volume during fasting and 32 min after a liquid nutritional supplement meal. Subjects reported to the clinic after an overnight fast. 99mTC was given by an intravenous injection in the forearm. The first fasting scan was obtained, and the study medication was given s.c. After 10 min, a 2nd fasting post medication scan was obtained, and the meal consumed; then two serial postprandial scans were obtained. Each scan required 9-12 min. Tomographic images of the gastric wall were obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content.
Time Frame: 16 weeks (approximately 1 hour after 99mTC injection)
Population: Intent to treat analysis; data were imputed for the 5 participants who dropped out.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 19 | 21
mL | 453 [378 to 536] | 433 [408 to 602]
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 17/19 | 14/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=19) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 12 (31) | 2 (5)
Bloating (Gastrointestinal disorders) | 2 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Headache (General disorders) | 5 (7) | 4 (5)
Abdominal pain/discomfort (Gastrointestinal disorders) | 4 (5) | 2 (3)
Abdominal Cramping (Gastrointestinal disorders) | 3 (4) | 2 (3)
Lightheaded (General disorders) | 1 (1) | 2 (2)
Loose stools (Gastrointestinal disorders) | 3 (3) | 1 (2)
Decreased appetite (Gastrointestinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes